CLINICAL TRIAL: NCT04790136
Title: Characterisation of Relative Bioavailability of GLA-015 in Comparison With an Oily Cannabidiol Solution (NRF 22.10) - a Multiple Dose, Randomised, 2-period Crossover-trial With Twice Daily Administration in Healthy Adult Male and Female Subjects
Brief Title: Cannabidiol Bioavailability Trial With Oral Multiple Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SocraTec R&D GmbH (Other)
Collaborators: Glatt Pharmaceutical Services GmbH & Co. KG (Unknown); SocraMetrics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1393cbd20ct; 2020-004807-15 (EudraCT Number)
Record Dates: First submitted 2021-03-03; First posted 2021-03-10 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Comparative Bioavailability
Keywords: Bioavailability; Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLA-015 (Experimental): GLA-015 (Glatt Pharmaceutical Services GmbH & Co. KG, Germany); 5.051 g granules containing 1500 mg cannabidiol to be dispersed in water; oral multiple dose administration twice daily over 7 consecutive days after a light meal
  Interventions: Drug: GLA-015
- DAC C-052 "Cannabidiol" / NRF 22.10 "Oily cannabidiol solution 100 mg/ml" (Active Comparator): DAC C-052 "Cannabidiol" / NRF 22.10 "Ölige Cannabidiol-Lösung 100 mg/ml" ("Oily cannabidiol solution 100 mg/ml") (Glatt Pharmaceutical Services GmbH & Co. KG, Germany; according to DAC/NRF specifications); 15 ml solution containing 1500 mg cannabidiol; oral multiple dose administration twice daily over 7 consecutive days after a light meal
  Interventions: Drug: DAC C-052 "Cannabidiol" / NRF 22.10 "Oily cannabidiol solution 100 mg/ml"

INTERVENTIONS:
Drug: GLA-015 — administration followed by PK blood sampling
  Arms: GLA-015
Drug: DAC C-052 "Cannabidiol" / NRF 22.10 "Oily cannabidiol solution 100 mg/ml" — administration followed by PK blood sampling
  Arms: DAC C-052 "Cannabidiol" / NRF 22.10 "Oily cannabidiol solution 100 mg/ml"

SUMMARY:
Glatt Pharmaceutical Services GmbH & Co. KG is developing a new CBD granules formulation (GLA-015 / Cannabidiol 1500 mg 29,7% w/w GRA BLD P) which is intended to be used in the treatment of the new Coronavirus disease 2019 (COVID-19). Due to its enhanced solubility the new product is expected to show increased bioavailability, reduced variability especially in the fasted state and better robustness towards food interaction compared to oil-based cannabidiol solutions.

The aim of the present clinical trial is the characterisation of maximum systemic exposure of CBD and its active metabolite 7-OH-CBD of the newly developed Test product in the estimated target effective dose for treatment of COVID-19 as well as the comparison of its systemic bioavailability to CBD administered as oily solution.

Comparison of maximum systemic exposure of Test vs. Reference will be performed under steady state conditions with twice daily intake after a light meal over 7 consecutive days.

DETAILED DESCRIPTION:
This single centre, open-label, randomised (order of treatments), balanced, multiple dose trial will be performed in a 2-period, 2-sequence-crossover design with direct switch-over. Eighteen (18) healthy subjects of both sexes (balanced distribution intended, but minimum 40% of each sex) are intended to be randomised.

The IMPs will be administered after a light meal as single oral doses of 1500 mg cannabidiol (i.e. 5.051 g granules of Test to be dispersed in water or 15 ml solution of Reference) twice daily (i.e. every 12 h) over 7 consecutive days.

Blood sampling will be performed after the 13th administration over 24 h, thereby including the 14th administration, in order to characterise pharmacokinetic parameters after multiple dosing over a whole day interval.

Comparison of maximum systemic exposure of Test vs. Reference will be performed under steady state conditions by means of AUC144-168,ss, Cmax,144-168,ss, and Cmin,144-168,ss of CBD and 7-OH-CBD.

The clinical trial will be performed as a cross-over investigation with intra-individual comparison, thus reducing variability of the pharmacokinetic parameters, which is supposed to be higher between subjects than within an individual subject.

ELIGIBILITY:
Inclusion Criteria:

1. ethnic origin: Caucasian
2. age: 18 years or older (including)
3. body-mass index (BMI): >= 18.5 kg/m² and <= 30.0 kg/m²
4. good state of health
5. non-smoker or ex-smoker for at least 1 month
6. written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical trial

Exclusion Criteria:

Safety concerns

1. existing cardiac and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient
2. existing hepatic and/or renal diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredient
3. existing gastrointestinal diseases or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient
4. history of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
5. hepatic impairment
6. history of bradycardia, tachycardia or other arrhythmic symptoms of clinical significance
7. Nurses Global Assessment of Suicide Risk (NGASR)-scale showing a high or very high risk
8. known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparations
9. history of severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the investigator
10. systolic blood pressure < 90 or > 139 mmHg
11. diastolic blood pressure < 60 or > 89 mmHg
12. heart rate < 50 bpm or > 90 bpm
13. QTc interval > 450 ms for men and > 470 ms for women
14. ASAT > 20% ULN, ALAT > 10% ULN, bilirubin > 20% ULN (except in case of existing Morbus Gilbert-Meulengracht deduced from anamnesis/medical history) and creatinine > 0.1 mg/dL ULN (limit of > 0.1 mg/dL correspondents to of > 9 µmol/l ULN)
15. all other laboratory values out of normal range unless the deviation from normal is judged as not relevant for the clinical trial by the investigator
16. positive anti-HIV-test (if positive to be verified by western blot), HBs-AG-test or anti-HCV-test
17. diagnosis of COVID-19 within the last 14 days prior to individual enrolment of the subject
18. contact to persons in foreign risk regions as defined by the Robert Koch Institute within the last 14 days prior to individual enrolment of the subject
19. known direct contact with insufficient protection to persons with diagnosis of COVID-19 within the last 14 days prior to individual enrolment upon reporting of the subject

    Lack of suitability for the clinical trial
20. acute or chronic diseases which may interfere with the pharmacokinetics of the IMP
21. history of or current drug or alcohol dependence
22. positive alcohol, cotinine or drug test at screening examination
23. regular intake of alcoholic food or beverages of ≥ 24 g pure ethanol for male or ≥ 12 g pure ethanol for female per day
24. subjects who are on a diet which could affect the pharmacokinetics of the active ingredient
25. regular intake of caffeine containing food or beverages of ≥ 500 mg caffeine per day
26. blood donation or other blood loss of more than 400 ml within the last 2 months prior to individual enrolment of the subject
27. administration of any investigational medicinal product during the last 2 months prior to individual enrolment of the subject
28. regular treatment with any systemically available medication (except hormonal contraceptives and hormonal replacement therapy, e.g. estrogens, L-thyroxine)
29. subjects, who report a frequent occurrence of migraine attacks

    For female subjects with childbearing potential only:
30. positive pregnancy test at screening examination
31. pregnant or lactating women
32. female subjects who do not agree to apply highly effective contraceptive methods

    Administrative reasons
33. subjects suspected or known not to follow instructions
34. subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Comparison of relative bioavailability of Test vs. Reference after multiple dose administration after a light meal determined by use of AUC144-168,ss of cannabidiol | 24 hours
  AUC144-168,ss = partial area under the concentration vs. time curve over both dosing intervals on PK profiling day (i.e. starting with the morning dose on study day 7 to 12 h after the evening dose on study day 7), calculated by means of the linear up/log down method (linear trapezoidal rule for increases in concentration/logarithmic trapezoidal rule for decreases in concentrations)
Comparison of relative bioavailability of Test vs. Reference after multiple dose administration after a light meal determined by use of Cmax,144-168,ss of cannabidiol | 24 hours
  Cmax,144-168,ss = observed maximum concentration over both dosing intervals on PK profiling day (i.e. starting with the morning dose on study day 7 to 12 h after the evening dose on study day 7), considering scheduled times
Comparison of relative bioavailability of Test vs. Reference after multiple dose administration after a light meal determined by use of Cmin,144-168,ss of cannabidiol | 24 hours
  Cmin,144-168,ss = (absolute) minimum concentrations over both dosing intervals on PK profiling day (i.e. starting with the morning dose on study day 7 to 12 h after the evening dose on study day 7), considering scheduled times
Comparison of relative bioavailability of Test vs. Reference after multiple dose administration after a light meal determined by use of AUC144-168,ss of 7-OH-CBD | 24 hours
  AUC144-168,ss = partial area under the concentration vs. time curve over both dosing intervals on PK profiling day (i.e. starting with the morning dose on study day 7 to 12 h after the evening dose on study day 7), calculated by means of the linear up/log down method (linear trapezoidal rule for increases in concentration/logarithmic trapezoidal rule for decreases in concentrations)
Comparison of relative bioavailability of Test vs. Reference after multiple dose administration after a light meal determined by use of Cmax,144-168,ss, of 7-OH-CBD | 24 hours
  Cmax,144-168,ss = observed maximum concentration over both dosing intervals on PK profiling day (i.e. starting with the morning dose on study day 7 to 12 h after the evening dose on study day 7), considering scheduled times
Comparison of relative bioavailability of Test vs. Reference after multiple dose administration after a light meal determined by use of Cmin,144-168,ss of 7-OH-CBD | 24 hours
  Cmin,144-168,ss = (absolute) minimum concentrations over both dosing intervals on PK profiling day (i.e. starting with the morning dose on study day 7 to 12 h after the evening dose on study day 7), considering scheduled times

SECONDARY OUTCOMES:
Frequency of Adverse Events | 14 days
  Descriptive statistics with regard to frequency of adverse events considering intensity, relationship to the IMP, action taken, outcome, and seriousness as well as period and treatment
Frequency of subjects showing Adverse Events | 14 days
  Descriptive statistics with regard to frequency of subjects showing adverse events considering intensity, relationship to the IMP, action taken, outcome, and seriousness as well as period and treatment

CONTACTS AND LOCATIONS:
Overall Officials: Frank Donath, Principal Investigator — SocraTec R&D GmbH Clinical Pharmacology Unit
Locations (1):
- SocraTec R&D GmbH Clinical Pharmacology Unit, Erfurt, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No